CLINICAL TRIAL: NCT06398197
Title: Nourish Pilot & CoDesign Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: American University (Other); Purdue University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20231429; CA2115405 (Other Grant/Funding Number: National Science Foundation)
Record Dates: First submitted 2024-04-26; First posted 2024-05-03 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Nutrition, Healthy
Keywords: Food Literacy; Cooking Skills
MeSH Terms: interventions — Cooking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment Group (Experimental): Subjects first participate in 8 weekly cooking classes immediately after baseline data collection ends.
  Interventions: Behavioral: cooking and food skills intervention
- Delayed intervention control group (No Intervention): Subjects receive no intervention for 9 weeks, serving as the control group. Once all data collection is complete, the delayed intervention control group will receive the intervention (8 weekly cooking classes)

INTERVENTIONS:
Behavioral: cooking and food skills intervention — Participants will attend a weekly in-person class with brief instructional video clips, hands-on cooking and tasting experiences. Participants will work individually and as part of small groups during instructional sessions. At the end of each class, participants will receive a grocery bundle and a kitchen gadget that serves both as an incentive and implementation support to promote improved cooking frequency and confidence. Participants will be asked to post photos of what they made with their groceries to an instant messaging software (GroupMe application) and be encouraged to engage with fellow classmates on GroupMe to encourage social support of cooking. The intervention ends after the 8, weekly classes conclude (8 weeks total intervention time)
  Other Names: Nourish
  Arms: Immediate Treatment Group

SUMMARY:
The purpose of the research study is to learn more about the best ways to teach cooking and food skills to adults, and how cooking classes may help reduce one's stress and food waste, as well as improve their diet.

DETAILED DESCRIPTION:
Currently, 12.8% of Americans experience food insecurity, and food insecurity is associated with elevated perceived stress. Food literacy is proficiency in food-related skills and knowledge, including food preparation and cooking skills, basic nutrition knowledge, and the ability to prevent food waste. Recent research conducted in Australia suggests that food literacy interventions are associated with improved food security. Traditionally food literacy interventions take a recipe-based approach to culinary nutrition and lack information about key components of food literacy, such as food storage and food waste reduction techniques. However, recent research by the PI contends that recipes may be difficult for food insecure individuals to implement at home, given the challenge of procuring ingredients, suggesting the need for a new approach. In addition, food insecure households face additional environmental challenges, such as owning fewer cooking utensils, compared to food secure households. Based on the Social Cognitive Theory, the Nourish intervention addresses these limitations by incorporating food waste reduction, food storage knowledge, and improvisational cooking skills (cooking with what you have on hand) into food literacy and culinary nutrition education, as well as providing key cooking utensils. Eventually, the study team plans to test the impact of the Nourish intervention on food literacy, perceived stress, diet quality and food security to determine if food literacy interventions can positively impact perceived stress, diet, and food security. The present pilot study will test the feasibility and acceptability of the Nourish intervention and corresponding evaluation, as well as provide participant feedback on the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Ability to attend classes in person

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Prescott, PhD, Principal Investigator — Case Western Reserve University; Brenna Ellison, PhD, Principal Investigator — Purdue University
Locations (1):
- Community Recruitment, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Within 20 minutes of participant informed consent, enrolled participants were randomized into groups. All enrolled participants were randomized.
Period: Overall Study
Arm/Group | Immediate Treatment Group | Delayed Intervention Control Group
Started | 18 | 8
Completed | 4 | 2
Not Completed | 14 | 6

BASELINE CHARACTERISTICS:
Population: There was missing data from 20 participants that could not be used in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment Group | Delayed Intervention Control Group | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Full Range); unit: Years] — Age in years
  Years | 38.25 [25 to 51] | 51.5 [46 to 57] | 42.67 [25 to 57]
Sex/Gender, Customized [Count of Participants; unit: Participants] — What is your Gender?
  Participants
    Male | 1 | 0 | 1
    Female | 3 | 2 | 5
    Other | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Food Waste Volume
Description: Food waste volume will be measured in grams using a study-provided food scale and waste log. Participants are asked to weigh discarded food and log the weight in a food waste tracking notebook for a period of 1 week prior to randomization at Baseline, and again for a period of 1 week at 10 weeks post-randomization. The outcome measure will use the difference in total volume of food waste between the two time points (post total food waste - pre total food waste).
Time Frame: Change from Baseline to 10 weeks post-randomization
Population: All participants that provided outcomes data were included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Immediate Treatment Group | Delayed Intervention Control Group
Number analyzed (Participants) | 4 | 2
grams | -796.19 (2231.81) | 2308.38 (452.37)

ADVERSE EVENTS:
Time Frame: From enrollment to follow-up, up to 20 weeks
Description: This study used the ClinicalTrials.gov definitions for adverse events.
Arm/Group | Immediate Treatment Group | Delayed Intervention Control Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/8
Other Adverse Events (participants affected / at risk) | 0/18 | 0/8

LIMITATIONS AND CAVEATS:
The primary outcome could not be analyzed for all participants. As a feasibility pilot, technical problems with measurement led to unreliable or uninterpretable data. In addition, there was a high amount of missing data. The small sample limits generalizability, and no conclusions about effectiveness can be drawn. Insights will guide methodological changes to reduce participant measurement burden and data collection errors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT06398197/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT06398197/ICF_000.pdf